CLINICAL TRIAL: NCT03680170
Title: The Effect of Home-based Working Memory Updating Training on Cognition and Health in Patients With Parkinson's Disease
Brief Title: Cognitive Training in Parkinson's Disease, the iPARK Study
Acronym: iPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: Karlstad University (Other)
Responsible Party: Principal Investigator, Anna Stigsdotter Neely, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: dnr 2014-1654; dnr 2017-02371 (Other Grant/Funding Number: The Swedish Research Council)
Record Dates: First submitted 2018-04-20; First posted 2018-09-21 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Cognitive Impairment
Keywords: Cognitive rehabilitation; Working memory; Randomized controlled trial; Placebo control
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two parallel assigned intervention groups with randomized allocation.The intervention of focus is a web-based working memory updating training. The placebo condition consists of a web-based low dose short term memory training. Both groups received pretesting (pre-test) before 30 sessions (6-8 weeks) of training followed by immediate post-testing (post-test 1) and a long term follow up four months after training (post-test 2)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: At the pre and first post test the person performing the testing is blinded to which group the participant is allocated to. The participant is blinded to which intervention he/she is participating in. At the second post-test the research assistant know which training the participant has been allocated to. Person performing the statistical analysis will be blinded to study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Working memory updating training (Experimental): Training with web-based program on the internet for 30 sessions (4-5 times a week). The result of the training is registered.
  Intervention Device: web-based cognitive training
  Interventions: Behavioral: Working memory updating training
- Placebo training (Placebo Comparator): Low dose, short term memory training. Intervention: Training with computer based program on the internet for 30 sessions (4-5 times a week).
  Intervention Device: Web-based cognitive training
  Interventions: Behavioral: Placebo training

INTERVENTIONS:
Behavioral: Working memory updating training — Each training session includes four working memory updating tasks that is performed at the participants home on their computer via internet. Each training session takes about 20 minutes to perform.
  Other Names: Web-based; Computer-based training; Internet-based training
  Arms: Working memory updating training
Behavioral: Placebo training — Each training session includes four short term memory tasks that is performed at the participants home on their computer via internet. Each training session takes about 20 minutes to perform.
  Other Names: Web-based training; Computer-based training; Internet-based training
  Arms: Placebo training

SUMMARY:
The aim of the iPARK-study is to investigate the effects of a process-based cognitive training program with focus on working memory in patients with Parkinson's Disease (PD). The study is a double blinded, randomized controlled trial with a parallel group design that aim to recruit 80 persons with PD. All patients will undergo 30 sessions (6-7 weeks) of web-based cognitive training performed at home. The working memory training is a process-based training program focusing specific on updating. The placebo program is a low dose short term memory paradigm without updating. A battery of neuropsychological tests (working memory, attention, episodic memory, inhibition control, risk taking and motoric speed) and questionnaires (everyday functioning and psychological health) will be performed before training and directly after training and after 16 weeks. Patient expectation and measures of adherence (motivation and results during training) will be controlled for.

The iPARK trial is expected to provide novel and clinical useful information whether updating training is an effective training paradigm in PD. Further it will hopefully contribute to a better understanding of cognitive function in PD.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is after Alzheimers disease (AD) the most common neurodegenerative disease with a prevalence of 1% of the population over 60 years of age. The cardinal symptoms are motoric and are believed to be caused by depletion of dopamine in the brain with severe depletion in the striatum. In addition to the motor impairments, there are several non-motor functions also affected, where cognitive decline and dementia are among the most common problems. Some claim that up to 75% of the total PD population will eventually develop dementia. Prior to dementia, milder cognitive problems are common and already at the time of diagnosis up to 42.5% of patients with PD are affected by decline in different cognitive functions. Early cognitive deficits seen is inhibition, shifting, working memory and planning, but a cognitive profile of visuospatial decline, semantic fluency and episodic memory has been connected to Parkinson's Disease Dementia (PDD). The occurrence of Lewy-bodies and Alzheimer type brain pathology is common in PDD but dopamine depletion has also been connected to cognitive decline in healthy elderly and in PD.

Although prescription of dementia medication in PD most likely has increased during the last decade there are limited evidence of treatment effects . This particular patient group is already burdened by polypharmacy and therefore investigating non-pharmacological interventions is of crucial importance. A recent systematic review of cognitive intervention studies in PD suggests that there is evidence of clinically meaningful improvements in overall cognition and moderate to large effect sizes on measures of working memory, processing speed and executive functions. Another review on the topic suggested that the results are promising, at least in the immediate or short term for some cognitive domains, but due to inconsistencies between studies and lack of methodological salience there are still a lot of questions unanswered. Baseline factors such as cognitive functioning, Hoehn and Yahr stage, premorbid intelligence all can have contributing effects on individual differences in training gain. Therefore it is important to thoroughly investigate baseline characteristics.

In the future, studies need to include more participants, be hypothesis driven and include more detail of the cognitive profile, training intervention and outcome measures.

One approach to cognitive training that has received a lot of attention and critique is process-based cognitive training, such as training focusing on working memory (WM) and executive functions (EF). The purpose of the process based approach is to strengthen general cognitive processes important to global cognitive functioning. WM and EF play central roles in several different functions such as episodic memory, reading comprehension and problem solving to mention a few. Research has also shown that WM and EF is negatively affected both in normal and pathological aging, such as PD.

Training of executive functioning and working memory have gained some promising results in healthy adults, showing improvements in working memory and executive functioning but there is also an indication of broader generalizations of training gain. Previously the effect of process-based updating training in healthy young and older individuals has been studied. Results showed that a period of updating training increased Blood Oxygen Level Dependent (BOLD) activity in striatum related to increased cognitive performance in both groups. Also a corresponding effect of training on dopaminergic neurotransmission was detected.

In the light of the dopamine dysfunction in PD, with negative effects on both motoric and cognitive function it is of interest to study if a non-invasive, non-pharmacological intervention can lead to better updating function with increased dopamine levels in patients with PD. The iPARK study is a double blinded randomized controlled trial that will examine the effect of a web-based cognitive training program with focus on updating training.

The primary question asked will be if updating training will improve the ability to update contents in working memory and also if there will be improvements in other cognitive functions such as psychomotor speed, working memory, executive functions and episodic memory. Further the aim is to investigate if there will be improvements in self-perceived everyday cognitive function and psychological health as well as if the effects seen will be sustained over a period of four months. Baseline factors will be investigated to see if they have a modulating effect on training. Further the iPARK trial will determine if a web-based training performed at home without active supervision is a feasible approach in this particular patient group. Compliance, adherence and expectations will be measured systematically.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's Disease according to United Kingdom Parkinson's Disease Brain Bank (UKPDSBB) criteria
2. Hoehn and Yahr stage I-III
3. Pathological dat scan
4. A score of 24 or over on the MMSE AND be without Dementia
5. Stable medication over the past three months
6. Owns and is able to use a home based computer or tablet with internet connection.

Exclusion Criteria:

1. Unstable medication
2. Ongoing cognitive training
3. Diagnosis of PDD
4. Drug or alcohol abuse

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Criterion task | 6-8 weeks (pretest-posttest 1)
  Improvement on Letter memory after 30 sessions of working memory training. total score:0-40 higher score indicate better performance total items:0-10 higher score indicate better performance
Criterion task | 16 weeks (posttest 1-posttest 2)
  Maintenance of Letter memory performance four months after completed working memory training.
  total score:0-40 higher score indicate better performance total items:0-10 higher score indicate better performance

SECONDARY OUTCOMES:
Transfer task n-back | 6-8 weeks (pretest-posttest 1)
  Improvement on updating performance measured by n-back (1,2 and 3 back) after 30 sessions of working memory training.
  1. back total score: 0-90 higher score indicate better performance
  2. back total score: 0-90 higher score indicate better performance
  3. back total score: 0-90 higher score indicate better performance
  1 back, Yes minus false alarms: 0-36 higher score indicate better performance 2 back, Yes minus false alarms: 0-36 higher score indicate better performance 3 back, Yes minus false alarms: 0-36 higher score indicate better performance
Transfer task n-back | 16 weeks (posttest 1-posttest 2)
  Maintenance of updating performance measured by n-back (1,2 and 3 back) four months after completed working memory training.
  1. back total score: 0-90 higher score indicate better performance
  2. back total score: 0-90 higher score indicate better performance
  3. back total score: 0-90 higher score indicate better performance
  1 back, Yes minus false alarms: 0-36 higher score indicate better performance 2 back, Yes minus false alarms: 0-36 higher score indicate better performance 3 back, Yes minus false alarms: 0-36 higher score indicate better performance
Transfer task digit memory running span | 6-8 weeks (pretest-posttest 1)
  Improvement on updating performance measured by digit memory running span after 30 sessions of working memory training.
  total score:0-40 higher score indicate better performance total items:0-10 higher score indicate better performance
Transfer task digit memory running span | 16 weeks (posttest 1-posttest 2)
  Maintenance of updating performance measured by digit memory running span four months after completed working memory training.
  total score:0-40 higher score indicate better performance total items:0-10 higher score indicate better performance
Updating total score | 6-8 weeks (pretest-posttest 1)
  Improvement in calculated composite score based on z-score((raw test score-mean of group)/standard deviation of group) for digit memory running span, 2-back and 3-back. Range -4 to 4. Higher z-score indicate better updating performance.
  (z score(3back yes-false alarms)+z score(2back yes-false alarms)+z score (digit memory running span total))/3
Updating total score | 16 weeks (posttest 1-posttest 2)
  Maintenance of calculated composite score based on z-score((raw test score-mean of group)/standard deviation of group) for digit memory running span, 2-back and 3-back. Range -4 to 4. Higher z-score indicate better updating performance.
  (z score(3back yes-false alarms)+z score(2back yes-false alarms)+z score (digit memory running span total))/3
Transfer task episodic memory | 6-8 weeks (pretest-posttest 1)
  Improvement on episodic memory performance measured by Buschke Selective Reminding Procedure after 30 sessions of working memory training.
  total score: 0-74 higher score indicate better performance list learning: 0-74 delayed score:0-18 higher score indicate better performance
Transfer task episodic memory | 16 weeks (posttest 1-posttest 2)
  Maintenance of on episodic memory performance measured by Buschke Selective Reminding Procedure four months after completed working memory training.
  total score: 0-74 higher score indicate better performance list learning: 0-74 higher score indicate better performance delayed score:0-18 higher score indicate better performance
Transfer task digit span | 6-8 weeks (pretest-posttest 1)
  Improvement on working memory performance measured by Digit span forward, backwards and sequencing (WAIS IV) after 30 sessions of working memory training.
  digit span forward total score: 0-16 higher score indicate better performance digit span backwards total score: 0-16 higher score indicate better performance digit span sequencing total score:0-16 higher score indicate better performance
Transfer task digit span | 16 weeks (posttest 1-posttest 2)
  Maintenance of working memory performance measured by Digit span forward, backwards and sequencing (WAIS IV) after 30 sessions of working memory training.
  digit span forward total score: 0-16 higher score indicate better performance digit span backwards total score: 0-16 higher score indicate better performance digit span sequencing total score:0-16 higher score indicate better performance
Transfer task visuospatial-span | 6-8 weeks (pretest-posttest 1)
  Maintenance of visuospatial working memory performance measured by visuospatial span task, 0-18 higher score indicate better performance
Transfer task visuospatial-span | 16 weeks (posttest 1-posttest 2)
  Maintenance of visuospatial working memory performance measured by visuospatial span task, total score 0-18 higher score indicate better performance
working memory total score | 6-8 weeks (pretest-posttest 1)
  Improvement in calculated composite score based on z-score((raw test score-mean of group)/standard deviation of group) from digit span forward, digit span backward, digit span sequencing and visuospatial span task, higher score indicate better performance Range -4 to 4.
  (z score(digit span forward)+z score(digit span backward)+z score (digit span sequencing)+z score (visuospatial span task))/4
working memory total score | 16 weeks (posttest 1-posttest 2)
  Maintenance in calculated composite score based on z-score((raw test score-mean of group)/standard deviation of group) from digit span forward, digit span backward, digit span sequencing and visuospatial span task, higher score indicate better performance. Range -4 to 4.
  (z score(digit span forward)+z score(digit span backward)+z score (digit span sequencing)+z score (visuospatial span task))/4
Transfer task Matrices (WAIS IV) | 6-8 weeks (pretest-posttest 1)
  Improvement on problem solving performance measured by Matrices (WAIS IV) after 30 sessions of working memory training.
  total score: 0-26, higher score indicate better performance
Transfer task Matrices (WAIS IV) | 16 weeks (posttest 1-posttest 2)
  Maintenance of problem solving performance measured by Matrices (WAIS IV) after 30 sessions of working memory training.
  total score: 0-26, higher score indicate better performance
Transfer task Digit symbol | 6-8 weeks (pretest-posttest 1)
  Improvement on mental and psychomotor speed measured by Digit symbol after 30 sessions of working memory training.
  total score: 0-135, higher score indicate better performance
Transfer task Digit symbol | 16 weeks (posttest 1-posttest 2)
  Maintenance of mental and psychomotor speed measured by Digit symbol four months after completed working memory training.
  total score: 0-135, higher score indicate better performance
Transfer task Perdue pegboard | 6-8 weeks (pretest-posttest 1)
  Improvement in calculated mental and psychomotor speed measured by Perdue pegboard after 30 sessions of working memory training.
  total score right hand: 0-24, higher score indicate better performance total score left hand: 0-24 higher score indicate better performance total score both hands: 0-24higher score indicate better performance
Transfer task Perdue pegboard | 16 weeks (posttest 1-posttest 2)
  Maintenance of mental and psychomotor speed measured by Perdue pegboard four months after completed working memory training.
  total score right hand: 0-24, higher score indicate better performance total score left hand: 0-24 higher score indicate better performance total score both hands: 0-24higher score indicate better performance
Mental and psychomotor speed total score | 6-8 weeks (pretest-posttest 1)
  Improvement in calculated composite score based on z-score((raw test score-mean of group)/standard deviation of group) for Digit symbol and Perdue pegboard after 30 sessions of working memory training. higher score indicate better performance (range -4 to 4).
  (z score(Perdue pegboard)+z score(digit symbol))/2
Mental and psychomotor speed total score | 16 weeks (posttest 1-posttest 2)
  Maintenance of calculated composite score based on z-score((raw test score-mean of group)/standard deviation of group) from Digit symbol and Perdue pegboard four months after completed working memory training. higher score indicate better performance. (range -4 to 4).
  (z score(Perdue pegboard)+z score(digit symbol))/2
Transfer task Stroop test | 6-8 weeks (pretest-posttest 1)
  Improvement of executive functions measured by Stroop test (DKEFS) after 30 sessions of working memory training.
  color naming 0-90 seconds less time indicate better performance word naming 0-90 seconds less time indicate better performance inhibition 0-90 seconds less time indicate better performance Inhibition cost total score:0-90 seconds, less inhibition cost indicate better performance
Transfer task Stroop test | 16 weeks (posttest 1-posttest 2)
  Maintenance of executive functions measured by Stroop test (DKEFS) four months after completed working memory training.
  color naming 0-90 seconds less time indicate better performance word naming 0-90 seconds less time indicate better performance inhibition 0-90 seconds less time indicate better performance Inhibition cost total score:0-90 seconds, less inhibition cost indicate better performance
Transfer task Trail Making Test | 6-8 weeks (pretest-posttest 1)
  Improvement on executive functions measured by Trail Making Test A and B (DKEFS) after 30 sessions of working memory training.
  TMT A 0-250 seconds less time indicate better performance TMT B 0-350 seconds less time indicate better performance Shift cost (TMTB-TMTA): 0-200 seconds, less shift cost indicate better performance
Transfer task Trail Making Test | 16 weeks (posttest 1-posttest 2)
  Maintenance of executive functions measured by Trail Making Test A and B (DKEFS) four months after completed working memory training.
  TMT A 0-250 seconds less time indicate better performance TMT B 0-350 seconds less time indicate better performance Shift cost (TMTB-TMTA): 0-200 seconds, less shift cost indicate better performance
Executive function total score | 6-8 weeks (pretest-posttest 1)
  Improvement calculated composite score based on z-score((raw test score-mean of group)/standard deviation of group) of Stroop test and Trail Making Test A and B after 30 sessions of working memory training higher score indicate better performance. Range -4 to 4.
  (z score(-TMTB-TMTA)+z score(-inhibition cost))/2
Executive function total score | 16 weeks (posttest 1-posttest 2)
  Maintenance of calculated z-score ((raw test score-mean of group)/standard deviation of group) of Stroop test and Trail Making Test A and B after 30 sessions of working memory training higher score indicate better performance. Range -4 to 4.
  (z score(-TMTB-TMTA)+z score(-inhibition cost))/2
Transfer task subjective cognitive complaints | 6-8 weeks (pretest-posttest 1)
  Improvement on subjective memory complaints measured by Prospective retrospective memory questionaire after 30 sessions of working memory training.
  total score: 16-80 higher scores indicate more cognitive complaints prospective score: 0-100 higher scores indicate more cognitive complaints retrospective score: 0-100 higher scores indicate more cognitive complaints short term score: 0-100 higher scores indicate more cognitive complaints long term score: 0-100 higher scores indicate more cognitive complaints self cued score: 0-100 higher scores indicate more cognitive complaints environmentally cued: 0-100 higher scores indicate more cognitive complaints
Transfer task subjective cognitive complaints | 16 weeks (posttest 1-posttest 2)
  Maintenance of subjective memory complaints measured by Prospective retrospective memory questionaire four months after completed working memory training.total score: 16-80 higher scores indicate more cognitive complaints prospective score: 0-100 higher scores indicate more cognitive complaints retrospective score: 0-100 higher scores indicate more cognitive complaints short term score: 0-100 higher scores indicate more cognitive complaints long term score: 0-100 higher scores indicate more cognitive complaints self cued score: 0-100 higher scores indicate more cognitive complaints environmentally cued: 0-100 higher scores indicate more cognitive complaints

OTHER OUTCOMES:
Hospital Anxiety Depression scale (Depression and anxiety) | 6-8 weeks (pretest- posttest 1) 16 weeks (posttest 1 - posttest 2)
  Severity of depression and anxiety symptoms measured by Hospital Anxiety Depression scale Anxiety score: 0-21 higher score indicate more anxiety Depression score: 0-21 higher score indicate more depression
Short Form Health Survey sf-36 (Health status) | 6-8 weeks (pretest- posttest 1) 16 weeks (posttest 1 - posttest 2)
  Health status measured by the Short Form Health Survey (sf-36) physical functioning score: 0-100 higher scores indicate less problems role limitations score: 0-100 higher scores indicate less problems energy fatigue score: 0-100 higher scores indicate less problems emotional well being score: 0-100 higher scores indicate less problems social functioning score: 0-100 higher scores indicate less problems pain score: 0-100 higher scores indicate less problems general health: 0-100 higher scores indicate less problems
Short version of the Karolinska Sleep Questionnaire (Sleep status) | 6-8 weeks (pretest- posttest 1) 16 weeks (posttest 1 - posttest 2)
  Sleep status measured by the Short version of the Karolinska Sleep Questionnaire total score: 5-30 higher scores indicate better sleep
Parkinson's Disease Questionnaire PDQ-39 (Function and well being) | 6-8 weeks (pretest- posttest 1) 16 weeks (posttest 1 - posttest 2)
  Function and well being measured by Parkinson's Disease Questionnaire-39 (PDQ39) Mobility score: 0-100 higher scores indicate more problems Activity of Daily Living score: 0-100 higher scores indicate more problems Emotional well being score: 0-100 higher scores indicate more problems Stigma score: 0-100 higher scores indicate more problems Social support score: 0-100 higher scores indicate more problems Cognition score: 0-100 higher scores indicate more problems Communication score: 0-100 higher scores indicate more problems Bodily discomfort score: 0-100 higher scores indicate more problems Summary index: 0-100 higher scores indicate more problems
Urgency, Premeditation, Perseverance and Sensation Seeking Questionnaire UPPS (Impulsivity and risk taking) | 6-8 weeks (pretest- posttest 1) 16 weeks (posttest 1 - posttest 2)
  Impulsivity and risk taking measured by Urgency, Premeditation, Perseverance and Sensation Seeking Questionnaire (UPPS) Urgency score: 0-100 higher score indicate more urgency Premeditation score:0-100 higher score indicate less premeditation Perseverance score: 0-100 higher score indicate less perseverance Sensation seeking score: 0-100 higher score indicate more sensation seeking.
Balloon Analogue Risk Taking Task BART (Impulsivity and risk taking) | 6-8 weeks (pretest- posttest 1) 16 weeks (posttest 1 - posttest 2)
  Impulsivity and risk taking measured by the Balloon Analogue Risk Taking Task (BART).
  Number of explosions: 0-30
Checklist Individual Strength Questionnaire CIS (Fatigue) | 6-8 weeks (pretest- posttest 1) 16 weeks (posttest 1 - posttest 2)
  Fatigue measured by Checklist Individual Strength Questionnaire (CIS) after 30 sessions of working memory training.
  total score: 20-140
Adherence (Task engagement) | 6-8 weeks (during training)
  Task engagement is measured by self assessed motivation to training and ability to stay focused during training measured before and after each training session.
Compliance (Finishing training within time frame) | 6-8 weeks (during training)
  Compliance is measured by number of participants finishing the training within time frame, 6-8 weeks.
Age | before training (pretest)
  Demographic characteristic: age at baseline
sex | before training (pretest)
  Demographic characteristic: sex
Educational level | before training (pretest)
  Demographic characteristic: educational level
Disease duration | before training (pretest)
  Demographic characteristic: disease duration
Disease stage | before training (pretest)
  Disease characteristic: disease stage (Hoehn and Yahr stage) Range 0-4
Levodopa Equivalent Dose (Medication for Parkinson's Disease) | 6-8 weeks (pretest- posttest 1) 16 weeks (posttest 1 - posttest 2)
  Medication use measured by Levodopa Equivalent Dose
Unified Parkinson's Disease Rating Scale (Motor symptoms) | before training (pretest)
  Motor symptoms assessed by the Unified Parkinson's Disease Rating Scale part 3 Total score:0-108 (higher scores indicate more motor symptoms)
Mini Mental State Examination (Global cognitive function) | before training (pretest)
  Global cognitive function measured by Mini Mental State Examination (MMSE) Total score: 24-30 (patients with lower scores is not included), lower scores indicate worse performance.
Side (left or right) most affected of Parkinson's Disease symptoms | before training (pretest)
  Disease characteristic: Most affected and starting side (Parkinsons symptoms)
Swedish vocabulary test SRB (Verbal ability) | before training (pretest)
  Verbal ability measured by Swedish vocabulary test (SRB). total score: 0-30 higher scores indicate better performance
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | 6-8 weeks (during training and at post test)
  All adverse events connected to training reported from participants and/or family members throughout the training period and after training are registered.

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Neely, Prof, Principal Investigator — Karlstad University
Locations (1):
- Umeå University department of psychology, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Background] de Lau LM, Breteler MM. Epidemiology of Parkinson's disease. Lancet Neurol. 2006 Jun;5(6):525-35. doi: 10.1016/S1474-4422(06)70471-9. PMID 16713924
- [Background] Aarsland D, Kurz MW. The epidemiology of dementia associated with Parkinson disease. J Neurol Sci. 2010 Feb 15;289(1-2):18-22. doi: 10.1016/j.jns.2009.08.034. Epub 2009 Sep 4. PMID 19733364
- [Background] Elgh E, Domellof M, Linder J, Edstrom M, Stenlund H, Forsgren L. Cognitive function in early Parkinson's disease: a population-based study. Eur J Neurol. 2009 Dec;16(12):1278-84. doi: 10.1111/j.1468-1331.2009.02707.x. Epub 2009 Jun 15. PMID 19538208
- [Background] Yarnall AJ, Breen DP, Duncan GW, Khoo TK, Coleman SY, Firbank MJ, Nombela C, Winder-Rhodes S, Evans JR, Rowe JB, Mollenhauer B, Kruse N, Hudson G, Chinnery PF, O'Brien JT, Robbins TW, Wesnes K, Brooks DJ, Barker RA, Burn DJ; ICICLE-PD Study Group. Characterizing mild cognitive impairment in incident Parkinson disease: the ICICLE-PD study. Neurology. 2014 Jan 28;82(4):308-16. doi: 10.1212/WNL.0000000000000066. Epub 2013 Dec 20. PMID 24363137
- [Background] Kehagia AA, Barker RA, Robbins TW. Neuropsychological and clinical heterogeneity of cognitive impairment and dementia in patients with Parkinson's disease. Lancet Neurol. 2010 Dec;9(12):1200-1213. doi: 10.1016/S1474-4422(10)70212-X. Epub 2010 Sep 27. PMID 20880750
- [Background] Landau SM, Lal R, O'Neil JP, Baker S, Jagust WJ. Striatal dopamine and working memory. Cereb Cortex. 2009 Feb;19(2):445-54. doi: 10.1093/cercor/bhn095. Epub 2008 Jun 11. PMID 18550595
- [Background] Ekman U, Eriksson J, Forsgren L, Mo SJ, Riklund K, Nyberg L. Functional brain activity and presynaptic dopamine uptake in patients with Parkinson's disease and mild cognitive impairment: a cross-sectional study. Lancet Neurol. 2012 Aug;11(8):679-87. doi: 10.1016/S1474-4422(12)70138-2. Epub 2012 Jun 27. PMID 22742929
- [Background] Ito K, Nagano-Saito A, Kato T, Arahata Y, Nakamura A, Kawasumi Y, Hatano K, Abe Y, Yamada T, Kachi T, Brooks DJ. Striatal and extrastriatal dysfunction in Parkinson's disease with dementia: a 6-[18F]fluoro-L-dopa PET study. Brain. 2002 Jun;125(Pt 6):1358-65. doi: 10.1093/brain/awf134. PMID 12023324
- [Background] Seppi K, Weintraub D, Coelho M, Perez-Lloret S, Fox SH, Katzenschlager R, Hametner EM, Poewe W, Rascol O, Goetz CG, Sampaio C. The Movement Disorder Society Evidence-Based Medicine Review Update: Treatments for the non-motor symptoms of Parkinson's disease. Mov Disord. 2011 Oct;26 Suppl 3(0 3):S42-80. doi: 10.1002/mds.23884. PMID 22021174
- [Background] Leung IH, Walton CC, Hallock H, Lewis SJ, Valenzuela M, Lampit A. Cognitive training in Parkinson disease: A systematic review and meta-analysis. Neurology. 2015 Nov 24;85(21):1843-51. doi: 10.1212/WNL.0000000000002145. Epub 2015 Oct 30. PMID 26519540
- [Background] Glizer D, MacDonald PA. Cognitive Training in Parkinson's Disease: A Review of Studies from 2000 to 2014. Parkinsons Dis. 2016;2016:9291713. doi: 10.1155/2016/9291713. Epub 2016 Sep 5. PMID 27688923
- [Background] Klingberg T. Training and plasticity of working memory. Trends Cogn Sci. 2010 Jul;14(7):317-24. doi: 10.1016/j.tics.2010.05.002. Epub 2010 Jun 16. PMID 20630350
- [Background] Morrison AB, Chein JM. Does working memory training work? The promise and challenges of enhancing cognition by training working memory. Psychon Bull Rev. 2011 Feb;18(1):46-60. doi: 10.3758/s13423-010-0034-0. PMID 21327348
- [Background] Shipstead Z, Redick TS, Engle RW. Is working memory training effective? Psychol Bull. 2012 Jul;138(4):628-654. doi: 10.1037/a0027473. Epub 2012 Mar 12. PMID 22409508
- [Background] Unsworth N, Engle RW. Simple and complex memory spans and their relation to fluid abilities: Evidence from list-length effects. Journal of Memory and Language 54(1): 68-80, 2006.
- [Background] Unsworth N, Engle RW. The nature of individual differences in working memory capacity: active maintenance in primary memory and controlled search from secondary memory. Psychol Rev. 2007 Jan;114(1):104-32. doi: 10.1037/0033-295X.114.1.104. PMID 17227183
- [Background] Gabrieli JDE, Singh J, Stebbins GT, & Goetz CG. Reduced working memory span in Parkinson's disease: Evidence for the role of frontostriatal system in working and strategic memory. Neuropsychology, 10(3): 322-332,1996.
- [Background] McCabe DP, Roediger HL, McDaniel MA, Balota DA, Hambrick DZ. The relationship between working memory capacity and executive functioning: evidence for a common executive attention construct. Neuropsychology. 2010 Mar;24(2):222-243. doi: 10.1037/a0017619. PMID 20230116
- [Background] Chein JM, Morrison AB. Expanding the mind's workspace: training and transfer effects with a complex working memory span task. Psychon Bull Rev. 2010 Apr;17(2):193-9. doi: 10.3758/PBR.17.2.193. PMID 20382919
- [Background] Dahlin E, Neely AS, Larsson A, Backman L, Nyberg L. Transfer of learning after updating training mediated by the striatum. Science. 2008 Jun 13;320(5882):1510-2. doi: 10.1126/science.1155466. PMID 18556560
- [Background] Backman L, Nyberg L, Soveri A, Johansson J, Andersson M, Dahlin E, Neely AS, Virta J, Laine M, Rinne JO. Effects of working-memory training on striatal dopamine release. Science. 2011 Aug 5;333(6043):718. doi: 10.1126/science.1204978. PMID 21817043
- [Background] Dahlin E, Nyberg L, Backman L, Neely AS. Plasticity of executive functioning in young and older adults: immediate training gains, transfer, and long-term maintenance. Psychol Aging. 2008 Dec;23(4):720-30. doi: 10.1037/a0014296. PMID 19140643
- [Background] Backman L, Waris O, Johansson J, Andersson M, Rinne JO, Alakurtti K, Soveri A, Laine M, Nyberg L. Increased dopamine release after working-memory updating training: Neurochemical correlates of transfer. Sci Rep. 2017 Aug 2;7(1):7160. doi: 10.1038/s41598-017-07577-y. PMID 28769095
- [Derived] Walton L, Neely AS, Backstrom D, Eriksson Domellof M. The experience of process-based cognitive training in people with Parkinson's disease: a route to transfer to everyday life. Neuropsychol Rehabil. 2026 Feb 10:1-20. doi: 10.1080/09602011.2026.2613961. Online ahead of print. PMID 41667390
- [Derived] Domellof ME, Walton L, Boraxbekk CJ, Backstrom D, Josefsson M, Forsgren L, Stigsdotter Neely A. Evaluating a frontostriatal working-memory updating-training paradigm in Parkinson's disease: the iPARK trial, a double-blinded randomized controlled trial. BMC Neurol. 2020 Sep 7;20(1):337. doi: 10.1186/s12883-020-01893-z. PMID 32894075